CLINICAL TRIAL: NCT04993807
Title: Data-driven Shared Decision-Making (SDM) to Reduce Symptom Burden in Atrial Fibrillation (AF)
Brief Title: Data-driven SDM to Reduce Symptom Burden in AF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Meghan Turchioe, Assistant Professor of Nursing, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AAAU2028; K99NR019124 (NIH); 19-11021059 (Other: Weill Cornell Medicine)
Record Dates: First submitted 2021-07-27; First posted 2021-08-06 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation; Patient Engagement
Keywords: Shared Decision-Making (SDM); Symptom Burden; Decisional Conflict; Decision Regret; Decision Satisfaction
MeSH Terms: conditions — Atrial Fibrillation; Patient Participation

STUDY DESIGN:
Intervention Model Description: This is a single arm feasibility study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Shared decision-making tool (Experimental): Participants in this arm will view a shared decision-making tool while they are undergoing consultation to have an atrial fibrillation ablation.
  Interventions: Other: Shared decision-making tool

INTERVENTIONS:
Other: Shared decision-making tool — Participants will use an interactive web page intended to aid patient decision-making (i.e., a decision aid) while undergoing consultation for atrial fibrillation ablation.

SUMMARY:
This study is a single-group feasibility study evaluating decision aid visualizations which display common post-ablation symptom patterns as a tool for shared decision-making. The specific aim of the clinical trial is to evaluate the feasibility of putting the visualizations into clinical practice (n=75). The hypothesis is that patients will report low decisional conflict and decision regret and high satisfaction with their decision about whether to undergo an ablation or not.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common heart rhythm disorder, and nearly 90% of patients experience symptoms such as shortness of breath that directly impair their health-related quality of life (HRQoL). Catheter ablation is a minimally invasive, surgical procedure that is routinely performed to treat AF and associated symptoms with the goal of improving HRQOL, but also carries potentially serious risks. Shared decision-making (SDM), in which treatment decisions are aligned based on high quality evidence and patient values and goals of care, is a widely encouraged practice for navigating complex healthcare decisions such as these. However, SDM around rhythm and symptom management does not routinely occur due to a lack of detailed evidence about symptom improvement post-ablation, and a lack of decision aids to communicate evidence to patients. The overarching goal of this award is to create an interactive patient decision aid composed of established evidence from clinical trials together with novel "real world" evidence about symptom improvement post ablation mined from electronic health records (EHRs).

The investigators propose to use "real-world evidence" drawn from electronic health records (EHRs) to characterize post-ablation symptom patterns, and display them in decision-aid visualizations to support shared decision-making (SDM). In this project, the investigators will first use natural language processing (NLP) and machine learning (ML) to extract and analyze symptom data from narrative notes in EHRs. The investigators will also employ a rigorous, user-centered design protocol created during the Principal Investigator's post-doctoral work to develop decision-aid visualizations. In the clinical trial, the investigators will evaluate the feasibility of implementing these interactive decision-aid visualizations in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of paroxysmal AF according to International Classification of Diseases, Tenth Revision (ICD-10)
* Scheduled consultation at NewYork-Presbyterian Hospital (NYP) to discuss catheter ablation
* Symptomatic AF at baseline
* Age 18 years and older
* Able to read and speak English
* Willing/able to provide informed consent

Exclusion Criteria:

* Asymptomatic AF
* Severe cognitive impairment
* Major psychiatric illness
* Concomitant terminal illness that would preclude participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-03-25 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Decisional conflict assessed using the Decisional Conflict Scale | Baseline
  Conflict about the decision to undergo atrial fibrillation will be assessed using the Decisional Conflict Scale on a scale of 0 (no decisional conflict) to 100 (extremely high decisional conflict).
Decision regret assessed using the Decisional Regret Scale | 12 weeks
  Regret about the decision to undergo atrial fibrillation will be assessed using the Decision Regret Scale on a scale of 0 (no decision regret) to 100 (extremely high decision regret).
Decision satisfaction assessed using the Satisfaction with Decision Scale | 12 weeks
  Satisfaction about the decision to undergo atrial fibrillation will be assessed using the Satisfaction with Decision Scale on a scale of 1 (low satisfaction) to 5 (high satisfaction).

SECONDARY OUTCOMES:
Post-ablation symptom burden assessed using the Atrial Fibrillation severity Scale (AFSS) | 12 weeks
  The severity of atrial fibrillation symptoms after an ablation will be assessed using the AFSS on a scale of 0 (no symptom burden) to 35 (extremely high symptom burden).
Post-ablation health-related quality of life assessed using the Atrial Fibrillation Effect on QualiTy-of-Life (AFEQT) questionnaire | 12 weeks
  Health-related quality of life after an ablation will be assessed using the AFEQT on a scale of 0 (complete disability) to 100 (high quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Reading Turchioe, PhD, MPH, RN, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Weill Cornell Medicine, New York, New York
  - Columbia University Irving Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be available to other researchers upon reasonable request after Data Use Agreements have been executed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 years and ending 5 years following publication.
Access Criteria: Researchers who provide a methodologically sound proposal and have completed Data Use Agreements.